CLINICAL TRIAL: NCT03785782
Title: ARFI, VisR and DDAI Ultrasound for Improving Discrimination of Malignant and Unresponsive Breast Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1745
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Women scheduled for biopsy: 40 participants with diagnosed BIRADS-4a, 4b, 4c, or -5 masses will be recruited. The investigators aim to have approximately 10 in each of the BIRADS categories (4a, 4b, 4c, 5), resulting in 40 total subjects for Aim #1.
  Interventions: Device: Ultrasound
- Women scheduled for neoadjuvant chemo: 40 participants with malignant masses undergoing neoadjuvant chemotherapy (NAC) will be recruited.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Breast ultrasound

SUMMARY:
Purpose: The purpose of this study is to evaluate in vivo the diagnostic relevance of ultrasound-derived metrics for stiffness, elasticity, viscosity, and anisotropy.

Participants: Forty women with breast lesions that have a BIRADS-4 or BIRADS-5 rating and forty women undergoing neoadjuvant chemotherapy (NAC) for malignant breast lesions will be recruited. Subjects will be recruited from the Breast Imaging Division of UNC Hospitals.

Procedures (methods): In this exploratory clinical study, the investigators will attempt to demonstrate that ARFI, VisR, and DDAI ultrasound reliably detect malignant breast masses (Aim #1) and distinguish masses that respond to chemotherapy from those that do not (Aim #2). The ARFI, VisR, and DDAI imaging location will be on the surface of the breast, above the suspicious or malignant mass. This unblinded, open-label, exploratory study will be conducted in 40 women with diagnosed BIRADS-4 or -5 masses in Aim #1 and in 40 women with malignant masses undergoing neoadjuvant chemotherapy (NAC) in Aim #2.

DETAILED DESCRIPTION:
The primary objective of breast cancer screening is to identify early stage cancer, or precancerous lesions, at a time before symptoms emerge and when treatment is likely to result in a cure. Screening is beneficial when it averts progression of disease to metastasis and/or death, but adverse effects to patients (and unnecessary medical expense) may result downstream from false positives and indiscrimination of masses that will not respond to treatment. The sensitivity of digital mammography, the current screening standard in the US, has been reported in the range of 0.40 to 0.85, with a positive predictive value of 0.31. Sensitivity is increased by augmenting mammography with MRI and B-Mode ultrasound, but false positive rates may also increase3. There exists a vital need for a screening technology that exhibits high sensitivity and specificity for cancer detection with early identification of unresponsive masses.

This urgent need could be met by exploiting new imaging biomarkers. Specifically, the mechanical properties of breast tissue have been used for cancer detection, with both elasticity and viscosity demonstrated for discriminating malignant from benign lesions. Further, tissue anisotropy has been shown to correlate with core biopsy result and tumor grade, with large cancers significantly more anisotropic than small cancers. Importantly, while both MRI and ultrasound can be used to measure these biomarkers, ultrasound's cost effectiveness and ease of implementation render it an efficient platform to pursue.

The long-term goal of this research program is to develop a new ultrasound-based breast-screening tool to augment mammography. As a critical first step toward achieving this goal, the primary objective of the proposed research is to evaluate in vivo the diagnostic relevance of ultrasound-derived metrics for stiffness, elasticity, viscosity, and anisotropy. These biomarkers will be measured using novel, noninvasive ultrasound technologies under development in Dr. Gallippi's laboratory: 1) Acoustic Radiation Force Impulse (ARFI) ultrasound for interrogating tissue stiffness, 2) Viscoelastic Response (VisR) ultrasound for assessing tissue elasticity and viscosity, and 3) Dynamic Displacement Anisotropy Imaging (DDAI) for measuring tissue anisotropy. These technologies have been demonstrated previously for delineating atherosclerosis, muscular dystrophy, and renal dysfunction.

A.1.2.State the research question(s) (i.e., specific study aims and/or hypotheses).

The investigators hypothesize that ultrasound-derived stiffness, elasticity, viscosity, and anisotropy will correlate with lesion malignancy and response to treatment. To test this hypothesis, they will pursue the following specific aims:

Aim #1: Quantify the ability of ultrasound-derived stiffness, elasticity, viscosity, and anisotropy to detect malignancy. ARFI, VisR, and DDAI imaging will be performed on suspicious breast lesions in 40 women with BIRADS-4a, 4b, 4c, or -5 ratings. The diagnostic accuracy of imaging metrics will analyzed, with malignancy confirmed by histology as the outcome.

Aim #2: Quantify the ability of ultrasound-derived stiffness, elasticity, viscosity, and anisotropy to predict a positive response to treatment. ARFI, VisR, and DDAI imaging will be performed serially - once every four weeks over the course of neoadjuvant chemotherapy (NAC) - on malignant breast lesions in 40 women. Changes in outcome metrics over time will be correlated to overall reduction in tumor size (diameter and area). The ability of ultrasound metrics to predict a positive response to treatment will be examined. A positive response to treatment will be determined according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.

ELIGIBILITY:
Inclusion Criteria:

-

Aim 1:

Inclusion Criteria:

* Patients are 30-90 years of age
* Patients have breast masses with BIRADS 4a, 4b, 4c, or 5 rating
* Lesion is sonographically visible with B-Mode ultrasound on diagnostic workup
* Informed consent obtained and signed

Aim 2:

Inclusion Criteria:

* Patients are 30-90 years
* Patients who are or will be undergoing neoadjuvant chemotherapy (NAC) for stage 2 or 3 malignant breast lesions
* Lesion is sonographically visible with B-Mode ultrasound on diagnostic workup
* Informed consent is obtained and signed

Exclusion Criteria: Subjects who meet any of the exclusion criteria will be excluded from study participation for both Aim 1 and Aim 2.

* Inability to provide informed consent
* Inability to communicate in English
* Inability to remain motionless for 15 minutes
* Suspicious or malignant breast mass deeper than 3 cm from skin surface
* Previous biopsy or surgery to the site of the suspicious or malignant mass
* Patients who are pregnant
* Patients who are lactating
* Patients with a history of masectomy
* Patients with breast implants

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Study Population: Forty women with breast lesions that have a BIRADS-4 or BIRADS-5 rating and forty women undergoing neoadjuvant chemotherapy (NAC) for malignant breast lesions will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Gallippi, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Women Scheduled for Biopsy: Participants who have undergone breast ultrasonogram, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis.
- Women Scheduled for Neoadjuvant Chemo: Participants who have undergone breast ultrasonogram, malignant breast tumor was confirmed with biopsy and scheduled to receive neoadjuvant chemotherapy.
Period: Overall Study
Arm/Group | Women Scheduled for Biopsy | Women Scheduled for Neoadjuvant Chemo
Started | 40 | 5
Completed | 34 | 4
Not Completed | 6 | 1
Not completed — their lesions' were not suitable for the study criteria | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — insufficient image quality. | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women Scheduled for Biopsy | Women Scheduled for Neoadjuvant Chemo | Total
Number analyzed (Participants) | 39 | 5 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (14.0) | 54.4 (15.7) | 53.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 5 | 44
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 39 | 4 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 1 | 10
  White | 28 | 3 | 31
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 5 | 44

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Peak Displacement (PD) for Detecting Malignancy
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate peak displacement (PD) and correlated with biopsy findings of malignant or benign.
  Peak Displacement (PD) - Maximum displacement of tissue in the breast lesion after an Acoustic Radiation Force Impulse (ARFI) excitation.
  Participants who have undergone breast ultrasonogram were categorized as BIRADS-4a, 4b, 4c, or -5 masses.
Time Frame: Baseline imaging
Population: In total 34 subjects were included in the analysis. Six subjects were excluded because their lessons were unsuitable for the study criteria, had insufficient image quality, or were withdrawn. Biopsy finding of malignant:12 participants, Biopsy finding of benign: 22 participants. Women scheduled for neoadjuvant chemo are not included since they already have a malignant disease diagnosis.
Measure: Mean (Standard Error); unit: microns
Groups:
- Biopsy Finding of Malignant: Participants who have undergone breast ultrasonograms, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis. A biopsy was performed and cancer was confirmed.
- Biopsy Finding of Benign: Participants who have undergone breast ultrasonograms, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis. A biopsy was performed and cancer was not found.
Arm/Group | Biopsy Finding of Malignant | Biopsy Finding of Benign
Number analyzed (Participants) | 12 | 22
microns | 4.5803 (2.9947) | 8.628 (7.8776)
Statistical Analysis 1: Comparison: Biopsy Finding of Malignant; Test type: Other; p = 0.2988, Regression, Logistic

2. Primary Outcome: Weighted Correlation Between Peak Displacement (PD) to Predict Response to Neoadjuvant Chemotherapy.
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate peak displacement (PD) and correlated with biopsy findings of malignant or benign. Participants were imaged at baseline and end of each chemotherapy cycle. Patients were imaged 3-8 times w/ 3-4 weeks between scans.
  Peak Displacement (PD) - Maximum displacement of tissue in the breast lesion after an Acoustic Radiation Force Impulse (ARFI) excitation.
Time Frame: Up to 8 months
Population: Only women scheduled for neoadjuvant chemo and completed imaging (in total 4 subjects) were included in the analysis. One subject was withdrawn and was excluded from the analysis. Women scheduled for biopsy were not included.
Measure: Mean (Standard Error); unit: microns
Groups:
- Peak Displacement Before Neoadjuvant Chemo: peak displacement before neoadjuvant chemotherapy
- Peak Displacement After Neoadjuvant Chemo: peak displacement after neoadjuvant chemotherapy
Arm/Group | Peak Displacement Before Neoadjuvant Chemo | Peak Displacement After Neoadjuvant Chemo
Number analyzed (Participants) | 4 | 4
microns
  Responder to chemo: number analyzed (Participants) | 2 | 2
  Responder to chemo | 2.4715 (1.4746) | 6.7281 (3.5461)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2
  Non-responders to chemo | 2.5268 (1.3869) | 3.2511 (1.3869)
Statistical Analysis 1: Comparison: Peak Displacement Before Neoadjuvant Chemo vs Peak Displacement After Neoadjuvant Chemo; Test type: Other; p = 0.36, Regression, Linear

3. Primary Outcome: Weighted Correlation Between Displacement at a Given Time (TD) for ARFI to Predict Response to Neoadjuvant Chemotherapy
Description: The ultrasound data was processed to calculate displacement at a given time (TD) for ARFI and statistically correlated to response of treatment with neoadjuvant chemotherapy. These values were weighted based on the number of imaging visits during subjects' treatment. Acoustic Radiation Force Impulse (ARFI) - Ultrasound imaging technique in which a sacoustic pulse is transmitted into tissue, causing it to displace and recover in <1 ms. The tissue displacement was used to estimate stiffness and viscosity. Response to chemo - Defined as the lesion shrinking by 25% or more over the course of chemotherapy. Non-responders to chemo - Defined as lesion not shrinking by 25% or more over the course of chemotherapy. Participants were imaged at baseline and end of each chemotherapy cycle. Patients were imaged 3-8 times w/ 3-4 weeks between scans.
Time Frame: Up to 8 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: microns
Groups:
- Displacement at a Given Time (TD) for ARFI Before Neoadjuvant Chemo: displacement at a given time (TD) for ARFI before neoadjuvant chemo therapy
- Displacement at a Given Time (TD) for ARFI After Neoadjuvant Chemo: displacement at a given time (TD) for ARFI after neoadjuvant chemotherapy
Arm/Group | Displacement at a Given Time (TD) for ARFI Before Neoadjuvant Chemo | Displacement at a Given Time (TD) for ARFI After Neoadjuvant Chemo
Number analyzed (Participants) | 4 | 4
microns
  Responder to chemo: number analyzed (Participants) | 2 | 2
  Responder to chemo | 2.3495 (1.3904) | 6.1222 (3.0388)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2
  Non-responders to chemo | 2.2757 (1.1146) | 3.0156 (1.2928)
Statistical Analysis 1: Comparison: Displacement at a Given Time (TD) for ARFI Before Neoadjuvant Chemo vs Displacement at a Given Time (TD) for ARFI After Neoadjuvant Chemo; Test type: Other; p = 0.43, Regression, Linear

4. Primary Outcome: Weighted Correlation Between Relative Elasticity (RE) to Predict Response to Neoadjuvant Chemotherapy.
Description: The ultrasound data will be processed to calculate relative elasticity (RE) and statistically correlated to response of treatment with neoadjuvant chemotherapy. These values were weighted based on the number of imaging visits during subjects' treatment. Relative Elasticity (RE) - Qualitative estimate for tissue stiffness in the breast lesion based on VisR imaging. Response to chemo - Defined as the lesion shrinking by 25% or more over the course of chemotherapy. Non-responders to chemo - Defined as lesion not shrinking by 25% or more over the course of chemotherapy. Participants were imaged at baseline and end of each chemotherapy cycle. Patients were imaged 3-8 times w/ 3-4 weeks between scans.
Time Frame: Up to 8 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: 1/millimeter
Groups:
- Relative Elasticity Before Neoadjuvant Chemo: Relative Elasticity before neoadjuvant chemo therapy
- Relative Elasticity After Neoadjuvant Chemo: Relative Elasticity after neoadjuvant chemotherapy
Arm/Group | Relative Elasticity Before Neoadjuvant Chemo | Relative Elasticity After Neoadjuvant Chemo
Number analyzed (Participants) | 4 | 4
1/millimeter
  Responder to chemo: number analyzed (Participants) | 2 | 2
  Responder to chemo | 177.69 (69.91) | 89.41 (87.51)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2
  Non-responders to chemo | 190.51 (43.58) | 164.42 (87.51)
Statistical Analysis 1: Comparison: Relative Elasticity Before Neoadjuvant Chemo vs Relative Elasticity After Neoadjuvant Chemo; Test type: Other; p = 0.42, Regression, Linear

5. Primary Outcome: Weighted Correlation Between Relative Viscosity (RV) to Predict Response to Neoadjuvant Chemotherapy.
Description: The ultrasound data will be processed to calculate relative viscosity (RV) and statistically correlated to response of treatment with neoadjuvant chemotherapy. These values were weighted based on the number of imaging visits during subjects' treatment. Relative Viscosity (RV) - Qualitative estimate for tissue viscosity in the breast lesion based on VisR imaging. Response to chemo - Defined as the lesion shrinking by 25% or more over the course of chemotherapy. Non-responders to chemo - Defined as lesions not shrinking by 25% or more over the course of chemotherapy. Participants were imaged at baseline and end of each chemotherapy cycle. Patients were imaged 3-8 times w/ 3-4 weeks between scans.
Time Frame: Up to 8 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: milli second /millimeter
Groups:
- Relative Viscosity (RV) Before Neoadjuvant Chemo: Relative viscosity (RV) before neoadjuvant chemotherapy
- Relative Viscosity (RV) After Neoadjuvant Chemo: Relative viscosity (RV) after neoadjuvant chemotherapy
Arm/Group | Relative Viscosity (RV) Before Neoadjuvant Chemo | Relative Viscosity (RV) After Neoadjuvant Chemo
Number analyzed (Participants) | 4 | 4
milli second /millimeter
  Responder to chemo: number analyzed (Participants) | 2 | 2
  Responder to chemo | 384.55 (207.70) | 164.12 (85.79)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2
  Non-responders to chemo | 362.58 (179.51) | 281.54 (100.05)
Statistical Analysis 1: Comparison: Relative Viscosity (RV) Before Neoadjuvant Chemo vs Relative Viscosity (RV) After Neoadjuvant Chemo; Test type: Other; p = 0.45, Regression, Linear

6. Primary Outcome: Weighted Correlation Between Tissue Mass (TM) for VisR to Predict Response to Neoadjuvant Chemotherapy.
Description: The ultrasound data will be processed to calculate tissue mass (TM) for VisR and statistically correlated to the response of treatment with neoadjuvant chemotherapy. These values were weighted based on the number of imaging visits during subjects' treatment. Tissue Mass (TM) - Qualitative estimate for tissue mass in the breast lesion based on VisR imaging. Viscoelastic Response (VisR) - Ultrasound imaging technique in which a strong acoustic pulse is transmitted into the tissue, causing it to displace and recover. The tissue recovery curve is then fit to a mass-spring-damper physics model to estimate stiffness and viscosity. Response to chemo - Defined as the lesion shrinking by 25% or more over the course of chemotherapy. Non-responders to chemo - Defined as lesions not shrinking by 25% or more over the course of chemotherapy. Participants were imaged at baseline and end of each chemotherapy cycle. Patients were imaged 3-8 times w/ 3-4 weeks between scans.
Time Frame: Up to 8 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Kg/m
Groups:
- Tissue Mass (TM) for VisR Before Neoadjuvant Chemo: Tissue Mass (TM) for VisR before neoadjuvant chemotherapy
- Tissue Mass (TM) for VisR After Neoadjuvant Chemo: Tissue Mass (TM) for VisR after neoadjuvant chemotherapy
Arm/Group | Tissue Mass (TM) for VisR Before Neoadjuvant Chemo | Tissue Mass (TM) for VisR After Neoadjuvant Chemo
Number analyzed (Participants) | 4 | 4
Kg/m
  Responder to chemo: number analyzed (Participants) | 2 | 2
  Responder to chemo | 0.02 (0.02) | 0.05 (0.02)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2
  Non-responders to chemo | 0.03 (0.01) | 0.05 (0.03)
Statistical Analysis 1: Comparison: Tissue Mass (TM) for VisR Before Neoadjuvant Chemo vs Tissue Mass (TM) for VisR After Neoadjuvant Chemo; Test type: Other; p = 0.18, Regression, Linear

7. Primary Outcome: Comparison of ARFI PD Values at 90o Versus 0o Transducer Orientations for DDAI to Predict Response to Neoadjuvant Chemotherapy.
Description: The ultrasound data will be processed to calculate the ratio of ARFI PD values at 90o versus 0 o transducer orientations for DDAI and statistically correlated to the response of treatment with neoadjuvant chemotherapy. These values were weighted based on the number of imaging visits during subjects' treatment. Acoustic Radiation Force Impulse (ARFI) - Ultrasound imaging technique in which a strong acoustic pulse is transmitted into the tissue, causing it to displace and recover in less than a millisecond. The tissue displacement can be tracked and used to estimate stiffness and viscosity. Peak Displacement (PD) - Maximum displacement of tissue in the breast lesion after an ARFI excitation. Response to chemo - Defined as the lesion shrinking by 25% or more over the course of chemotherapy. Non-responders to chemo - Defined as lesions not shrinking by 25% or more. Participants were imaged at baseline and end of each chemotherapy cycle. Patients were imaged 3-8 times w/ 3-4 weeks btwn.
Time Frame: Up to 8 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: unitless ratio
Groups:
- ARFI PD Before Neoadjuvant Chemo 90 Degree: ARFI PD measured at 90 degrees transducer angle before neoadjuvant chemotherapy
- ARFI PD Before Neoadjuvant Chemo 0 Degree: ARFI PD measured at 0 degree transducer angle before neoadjuvant chemotherapy
- ARFI PD After Neoadjuvant Chemo 90 Degrees: ARFI PD measured at 90 degrees transducer angle after neoadjuvant chemotherapy
- ARFI PD After Neoadjuvant Chemo 0 Degree: ARFI PD measured at 0 degree transducer angle after neoadjuvant chemotherapy
Arm/Group | ARFI PD Before Neoadjuvant Chemo 90 Degree | ARFI PD Before Neoadjuvant Chemo 0 Degree | ARFI PD After Neoadjuvant Chemo 90 Degrees | ARFI PD After Neoadjuvant Chemo 0 Degree
Number analyzed (Participants) | 4 | 4 | 4 | 4
unitless ratio
  Responder to chemo: number analyzed (Participants) | 2 | 2 | 2 | 2
  Responder to chemo | 3.56 (3.08) | 2.11 (1.29) | 7.99 (5.80) | 6.06 (4.27)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2 | 2 | 2
  Non-responders to chemo | 2.52 (1.13) | 2.11 (1.29) | 7.99 (5.80) | 2.68 (0.10)
Statistical Analysis 1: Comparison: ARFI PD Before Neoadjuvant Chemo 90 Degree vs ARFI PD Before Neoadjuvant Chemo 0 Degree vs ARFI PD After Neoadjuvant Chemo 90 Degrees vs ARFI PD After Neoadjuvant Chemo 0 Degree; Test type: Other; p = 0.78, Regression, Linear

8. Primary Outcome: Comparison of Ratio of ARFI PD Values at 90o Versus 0o Transducer Orientations for DDAI to Predict Response to Neoadjuvant Chemotherapy.
Description: The ultrasound data was processed to calculate ratio of VisR RE values at 90o versus 0o transducer orientations for DDAI and statistically correlated to response of treatment with neoadjuvant chemotherapy. Values were weighted based on the number of imaging visits during subjects' treatment. Participants were imaged at baseline and end of each chemo cycle. Patients were imaged 3-8 times w/ 3-4 weeks btwn scans.
  Viscoelastic Response (VisR) - Ultrasound technique in which an acoustic pulse is transmitted into the tissue, causing it to displace and recover. Tissue recovery is fit to a mass-spring-damper physics model to estimate stiffness and viscosity.
  Relative Elasticity (RE) - Qualitative estimate for tissue stiffness in the breast lesion based on VisR imaging.
  Response to chemo - Defined as the lesion shrinking by 25% or more over the course of chemotherapy.
  Non-responders to chemo - Defined as lesions not shrinking by 25% or more over the course of chemotherapy.
Time Frame: Up to 60 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: unitless ratio
Groups:
- VisR -RE Before Neoadjuvant Chemo 90 Degree: VisR -RE measured at 90 degrees transducer angle before neoadjuvant chemotherapy
- VisR -RE Before Neoadjuvant Chemo 0 Degree: VisR -RE measured at 0 degree transducer angle before neoadjuvant chemotherapy
- VisR -RE After Neoadjuvant Chemo 90 Degrees: VisR -RE measured at 90 degrees transducer angle after neoadjuvant chemotherapy
- VisR -RE After Neoadjuvant Chemo 0 Degree: VisR -RE measured at 0 degree transducer angle after neoadjuvant chemotherapy
Arm/Group | VisR -RE Before Neoadjuvant Chemo 90 Degree | VisR -RE Before Neoadjuvant Chemo 0 Degree | VisR -RE After Neoadjuvant Chemo 90 Degrees | VisR -RE After Neoadjuvant Chemo 0 Degree
Number analyzed (Participants) | 4 | 4 | 4 | 4
unitless ratio
  Responder to chemo: number analyzed (Participants) | 2 | 2 | 2 | 2
  Responder to chemo | 155.59 (164.03) | 170.15 (8.74) | 69.45 (33.08) | 107.00 (81.34)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2 | 2 | 2
  Non-responders to chemo | 179.02 (1.84) | 185.64 (83.47) | 172.82 (153.11) | 160.95 (16.97)
Statistical Analysis 1: Comparison: VisR -RE Before Neoadjuvant Chemo 90 Degree vs VisR -RE Before Neoadjuvant Chemo 0 Degree vs VisR -RE After Neoadjuvant Chemo 90 Degrees vs VisR -RE After Neoadjuvant Chemo 0 Degree; Test type: Other; p = 0.45, Regression, Linear

9. Primary Outcome: Weighted Correlation Between Ratio of RV Values at 90o Versus 0o Transducer Orientations for DDAI to Predict Response to Neoadjuvant Chemotherapy.
Description: The ultrasound data will be processed to calculate ratio of RV values at 90o versus 0o transducer orientations for DDAI and statistically correlated to response of treatment with neoadjuvant chemotherapy. These values were weighted based on the number of imaging visits during subjects' treatment. Participants were imaged at baseline and end of each chemotherapy cycle. Patients were imaged 3-8 times w/ 3-4 weeks between scans.
  Relative Viscosity (RV) - Qualitative estimate for tissue viscosity in the breast lesion based on VisR imaging.
  Response to chemo - Defined as the lesion shrinking by 25% or more over the course of chemotherapy.
  Non-responders to chemo - Defined as lesion not shrinking by 25% or more over the course of chemotherapy.
Time Frame: Up to 8 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: unitless ratio
Groups:
- VisR -RV Before Neoadjuvant Chemo 90 Degree: VisR -RV measured at 90 degrees transducer angle before neoadjuvant chemotherapy
- VisR -RV Before Neoadjuvant Chemo 0 Degree: VisR -RV measured at 0 degree transducer angle before neoadjuvant chemotherapy
- VisR -RV After Neoadjuvant Chemo 90 Degrees: VisR -RV measured at 90 degrees transducer angle after neoadjuvant chemotherapy
- VisR -RV After Neoadjuvant Chemo 0 Degree: VisR -RV measured at 0 degree transducer angle after neoadjuvant chemotherapy
Arm/Group | VisR -RV Before Neoadjuvant Chemo 90 Degree | VisR -RV Before Neoadjuvant Chemo 0 Degree | VisR -RV After Neoadjuvant Chemo 90 Degrees | VisR -RV After Neoadjuvant Chemo 0 Degree
Number analyzed (Participants) | 4 | 4 | 4 | 4
unitless ratio
  Responder to chemo: number analyzed (Participants) | 2 | 2 | 2 | 2
  Responder to chemo | 289.93 (353.30) | 386.65 (288.47) | 144.27 (115.12) | 191.86 (100.15)
  Non-responders to chemo: number analyzed (Participants) | 2 | 2 | 2 | 2
  Non-responders to chemo | 322.84 (159.66) | 332.70 (241.89) | 231.17 (103.83) | 336.71 (52.55)
Statistical Analysis 1: Comparison: VisR -RV Before Neoadjuvant Chemo 90 Degree vs VisR -RV Before Neoadjuvant Chemo 0 Degree vs VisR -RV After Neoadjuvant Chemo 90 Degrees vs VisR -RV After Neoadjuvant Chemo 0 Degree; Test type: Other; p = 0.34, Regression, Linear

10. Primary Outcome: Correlation of Displacement at a Given Time (TD) for Detecting Malignancy.
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate displacement at a given time (TD) for ARFI and correlated with biopsy findings of malignant or benign.
  Acoustic Radiation Force Impulse (ARFI) - Ultrasound imaging technique in which a strong acoustic pulse is transmitted into tissue, causing it to displace and recover in less than a millisecond. The tissue displacement can be tracked and used to estimate stiffness and viscosity.
  Participants were imaged at baseline.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: microns
Groups:
- Biopsy Finding of Malignant: Participants who have undergone breast ultrasonogram, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis.
- Biopsy Finding is Benign: Participants who have undergone breast ultrasonograms, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis. A biopsy was performed and cancer was not found.
Arm/Group | Biopsy Finding of Malignant | Biopsy Finding is Benign
Number analyzed (Participants) | 12 | 22
microns | 4.16 (2.76) | 7.15 (5.54)
Statistical Analysis 1: Comparison: Biopsy Finding of Malignant; Test type: Other; p = 0.7465, Regression, Logistic

11. Primary Outcome: Correlation of Relative Elasticity (RE) for Detecting Malignancy.
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate relative elasticity (RE) and correlated with biopsy finding of malignant or benign.
  Relative Elasticity (RE) - Qualitative estimate for tissue stiffness in the breast lesion based on VisR imaging.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: 1/millimeter
Groups:
- Biopsy Result of Malignant: Participants who have undergone breast ultrasonograms, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis. A biopsy was performed and cancer was confirmed.
- Biopsy Result of Benign: Participants who have undergone breast ultrasonograms, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis. A biopsy was performed and cancer was not found.
Arm/Group | Biopsy Result of Malignant | Biopsy Result of Benign
Number analyzed (Participants) | 12 | 22
1/millimeter | 125.59 (69.69) | 89.88 (76.04)
Statistical Analysis 1: Comparison: Biopsy Result of Malignant; Test type: Other; p = 0.0466, Regression, Logistic

12. Primary Outcome: Correlation of Relative Viscosity (RV) for Detecting Malignancy.
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate relative viscosity (RV) and correlated with biopsy findings of malignant or benign.
  Relative Viscosity (RV) - Qualitative estimate for tissue viscosity in the breast lesion based on VisR imaging. Participants were imaged according to their neoadjuvant chemotherapy schedule, at baseline and end of each chemotherapy type
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: s/m
Groups:
- Biopsy Finding Was Malignant: Participants who have undergone breast ultrasonogram, categorized BIRADS-4a, 4b, 4c, or -5 masses requiring biopsy for the disease diagnosis.
Arm/Group | Biopsy Finding Was Malignant | Biopsy Finding of Benign
Number analyzed (Participants) | 12 | 22
s/m | 194.43 (170.13) | 137.60 (116.95)
Statistical Analysis 1: Comparison: Biopsy Finding Was Malignant; Test type: Other; p = 0.1567, Regression, Logistic

13. Primary Outcome: Correlation of Tissue Mass (TM) for VisR for Detecting Malignancy
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate tissue mass (TM) for VisRand correlated with biopsy findings of malignant or benign. Participants were imaged according to their neoadjuvant chemotherapy schedule, at baseline and end of each chemotherapy type Viscoelastic Response (VisR) - Ultrasound imaging technique in which a strong acoustic pulse is transmitted into the tissue, causing it to displace and recover. The tissue recovery curve is then fit to a mass-spring-damper physics model to estimate stiffness and viscosity.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Kg/m
Arm/Group | Biopsy Finding of Malignant | Biopsy Finding of Benign
Number analyzed (Participants) | 12 | 22
Kg/m | 0.46 (0.50) | 0.34 (0.31)
Statistical Analysis 1: Comparison: Biopsy Finding of Malignant; Test type: Other; p = 0.1837, Regression, Logistic

14. Primary Outcome: Correlation of Ratio of ARFI PD Values at 90o Versus 0o Transducer Orientations for Detecting Malignancy.
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate ratio of ARFI PD values at 90o versus 0o transducer orientations for DDAI and correlated with biopsy findings of malignant or benign. Participants were imaged according to their neoadjuvant chemotherapy schedule, at baseline and end of each chemotherapy type Acoustic Radiation Force Impulse (ARFI) - Ultrasound imaging technique in which a strong acoustic pulse is transmitted into the tissue, causing it to displace and recover in less than a millisecond. The tissue displacement can be tracked and used to estimate stiffness and viscosity.
  Peak Displacement (PD) - Maximum displacement of tissue in the breast lesion after an ARFI excitation.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: unitless ratio
Groups:
- ARFI PD 90 Degree: ARFI PD measured at 90 degrees transducer angle
- ARFI PD 0 Degree: ARFI PD measured at 0 degree transducer angle
Arm/Group | ARFI PD 90 Degree | ARFI PD 0 Degree
Number analyzed (Participants) | 34 | 34
unitless ratio
  Biopsy finding of malignant: number analyzed (Participants) | 12 | 12
  Biopsy finding of malignant | 4.88 (3.40) | 4.30 (2.45)
  Biopsy finding of benign: number analyzed (Participants) | 22 | 22
  Biopsy finding of benign | 9.84 (8.31) | 8.10 (7.34)
Statistical Analysis 1: Comparison: ARFI PD 90 Degree vs ARFI PD 0 Degree; Test type: Other; p = 0.7447, Regression, Logistic

15. Primary Outcome: Correlation of Ratio of VisR RE Values at 90o Versus 0o Transducer Orientations for Detecting Malignancy.
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate the ratio of VisR RE values at 90o versus 0o transducer orientations for DDAI and correlated with biopsy findings of malignant or benign. Participants were imaged according to their neoadjuvant chemotherapy schedule, at baseline and end of each chemotherapy type Viscoelastic Response (VisR) - Ultrasound imaging technique in which a strong acoustic pulse is transmitted into the tissue, causing it to displace and recover. The tissue recovery curve is then fit to a mass-spring-damper physics model to estimate stiffness and viscosity.
  Relative Elasticity (RE) - Qualitative estimate for tissue stiffness in the breast lesion based on VisR imaging.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: unitless ratio
Groups:
- VisR RE 90 Degree: VisR RE measured at 90 degrees transducer angle
- VisR RE 0 Degree: VisR RE measured at 0 degree transducer angle
Arm/Group | VisR RE 90 Degree | VisR RE 0 Degree
Number analyzed (Participants) | 34 | 34
unitless ratio
  Biopsy finding of malignant: number analyzed (Participants) | 12 | 12
  Biopsy finding of malignant | 139.66 (100.61) | 117.26 (70.72)
  Biopsy finding of benign: number analyzed (Participants) | 22 | 22
  Biopsy finding of benign | 77.47 (62.73) | 84.06 (74.92)
Statistical Analysis 1: Comparison: VisR RE 90 Degree vs VisR RE 0 Degree; Test type: Other; p = 0.0739, Regression, Logistic

16. Primary Outcome: Correlation of Ratio of VisR RV Values at 90o Versus 0o Transducer Orientations for Detecting Malignancy.
Description: The correlation of each ultrasound metric will be analyzed by constructing separate receiver operating characteristic (ROC) curves. The ultrasound data were processed to calculate ratio of VisR RV values at 90o versus 0o transducer orientations for DDAI and correlated with biopsy findings of malignant or benign. Participants were imaged according to their neoadjuvant chemotherapy schedule, at baseline and end of each chemotherapy type Displacement at Time (TD) - Displacement of tissue in the breast lesion at time t=0.2 ms after an ARFI excitation.
  Viscoelastic Response (VisR) - Ultrasound imaging technique in which a strong acoustic pulse is transmitted into tissue, causing it to displace and recover. The tissue recovery curve is then fit to a mass-spring-damper physics model to estimate stiffness and viscosity.
  Relative Viscosity (RV) - Qualitative estimate for tissue viscosity in the breast lesion based on VisR imaging.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: unitless ratio
Groups:
- VisR RV 90 Degree: VisR RV measured at 90 degrees transducer angle
- VisR RV 0 Degree: VisR RV measured at 0 degree transducer angle
Arm/Group | VisR RV 90 Degree | VisR RV 0 Degree
Number analyzed (Participants) | 34 | 34
unitless ratio
  Biopsy finding of malignant: number analyzed (Participants) | 12 | 12
  Biopsy finding of malignant | 161.10 (149.28) | 205.46 (132.67)
  Biopsy finding of benign: number analyzed (Participants) | 22 | 22
  Biopsy finding of benign | 113.67 (84.38) | 157.49 (142.23)
Statistical Analysis 1: Comparison: VisR RV 90 Degree vs VisR RV 0 Degree; Test type: Other; p = 0.9995, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Adverse events related to the imaging were collected directly following imaging for subjects in Arm 1. Adverse events were collected during the entire period where subjects were followed for Arm 2, which is up to 70 days.
Arm/Group | Women Scheduled for Biopsy | Women Scheduled for Neoadjuvant Chemo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/5
Other Adverse Events (participants affected / at risk) | 0/39 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT03785782/Prot_SAP_000.pdf
  • Informed Consent Form: Arm 1 (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT03785782/ICF_001.pdf
  • Informed Consent Form: Arm 2 (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT03785782/ICF_002.pdf